CLINICAL TRIAL: NCT05701566
Title: Use of Virtual Reality Technology as a Sedation Replacement During Colonoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 8177-21-IV-CTIL
Record Dates: First submitted 2023-01-18; First posted 2023-01-27 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-01

CONDITIONS: Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction | interventions — Colonoscopy

STUDY DESIGN:
Intervention Model Description: pilot randomized controled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual reality group (Experimental): unsedated colonoscopy using virtual reality headset.
  Interventions: Device: virtual reality headset
- colonoscopy with standard sedation (Active Comparator): standard sedated colonoscopy.
  Interventions: Other: colonoscopy with standard sedation.

INTERVENTIONS:
Device: virtual reality headset — use of virtual reality headset during colonoscopy as a substitute to sedation.
  Arms: virtual reality group
Other: colonoscopy with standard sedation. — use of standard sedation during colonoscopy.
  Arms: colonoscopy with standard sedation

SUMMARY:
A pilot non-randomized controlled study examined whether the use of VR technology can serve as an appropriate substitute for sedation in a colonoscopy examination.

DETAILED DESCRIPTION:
VR is an attention-distracting technology via visual and auditory signals by a computer-generated virtual engulfing environment. This technology has already been used in a variety of medical conditions and previous studies have demonstrated the benefit of using it as an additional tool for pain relief and as a substitute to sedation in invasive procedure. In this study we examined the use of VR as a substitute for sedation in colonoscopy. In this randomized control study, 60 patients were sequentially enrolled in a 1:1 ratio to either standard sedated colonoscopy or VR-unsedated procedure. The primary outcome was the overall satisfaction of patients who underwent unsedated colonoscopy with VR headset compared with patients who underwent standard sedation colonoscopy. Pain during the procedure, PDR, colonoscopy duration, post colonoscopy adverse events, post colonoscopy recovery and time-to-return to daily functions and turnaround time at the endoscopy unit were secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (≥18) with any elective indication for colonoscopy.

Exclusion Criteria:

* known seizures' disorders, cognitive, visual or auditory impairment.
* patients who were unable or unwilling to sign an informed consent.
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall satisfaction of patients who underwent un-sedated colonoscopy with virtual reality (VR) headset compared with patients who underwent standard sedation colonoscopy. | 1 day
  Questionnaire (1 - not satisfied at all, 5 - very satisfied)

SECONDARY OUTCOMES:
Pain during the procedure | 1 day
  Questionnaire (1- severe pain, 5 - no pain at all)
polyp detection rate (PDR) | during colonoscopy procedure
  number of polyps detected during colonoscopy
Colonoscopy duration | during colonoscopy procedure
  in minutes starting at insertion of the colonoscope to the anus until final withdrawal
Post colonoscopy adverse events | 1 day
  Questionnaire: Did you suffer from a general bad feeling after the test, including dizziness, nausea, abdominal pain (1 - no complaints at all, 5 - serious complaints)
Time-to-return to daily activities (work, driving) | 1 day
  hours
Turn-around time at the endoscopy Unit (overall duration of stay at the Endoscopy unit) | 1 day
  overall time at the unit

CONTACTS AND LOCATIONS:
Overall Officials: Ido Veisman, Dr., Principal Investigator — Sheba Medical Center
Locations (1):
- Gastroenterology department, Sheba Medical Center, Tel Litwinsky, Israel

IPD SHARING:
Plan to Share IPD: Undecided